CLINICAL TRIAL: NCT06368869
Title: The Effect of Different Types of Resin Cements on the Color Stability of Two Different Types of Ceramic Veneers (Randomized Controlled Clinical Trial)
Brief Title: The Effect of Different Types of Resin Cements on the Color Stability of Two Different Types of Ceramic Veneers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: amr elshimy (Other)
Responsible Party: Sponsor-Investigator, amr elshimy, Assistant Lecturer of Fixed Prosthodontics, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: #1/2022
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Color; Change Teeth, Posteruptive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Livento press veneers luted with dual cured resin cement (Experimental)
  Interventions: Other: Livento press veneers luted with dual cured resin cement
- Livento press veneers luted with light cured resin cement (Active Comparator)
  Interventions: Other: Livento press veneers luted with light cured resin cement
- Celtra duo veneers luted with dual cured resin cement (Experimental)
  Interventions: Other: Celtra duo veneers luted with dual cured resin cement
- Celtra duo veneers luted with light cured resin cement (Active Comparator)
  Interventions: Other: Celtra duo veneers luted with light cured resin cement

INTERVENTIONS:
Other: Livento press veneers luted with dual cured resin cement — Veneers will be fabricated using Lithium disilicate (Livento® Press) ceramic and luted using Bifix QM dual cured cement
  Arms: Livento press veneers luted with dual cured resin cement
Other: Livento press veneers luted with light cured resin cement — Veneers will be fabricated using Lithium disilicate (Livento® Press) ceramic and luted using Bisco choice 2 light cured cement
  Arms: Livento press veneers luted with light cured resin cement
Other: Celtra duo veneers luted with dual cured resin cement — Veneers will be fabricated using Zirconia-reinforced lithium silicate (Celtra® Press) ceramic and luted using Bifix QM dual cured cement
  Arms: Celtra duo veneers luted with dual cured resin cement
Other: Celtra duo veneers luted with light cured resin cement — Veneers will be fabricated using Zirconia-reinforced lithium silicate (Celtra® Press) ceramic and luted Bisco choice 2 light cured cement
  Arms: Celtra duo veneers luted with light cured resin cement

SUMMARY:
Aim of the study was to evaluate the color stability of lithium disilicate ceramic veneers and zirconia reinforced lithium silicate ceramic veneers by using two different types of resin cements including light cured and dual cured cements.

ELIGIBILITY:
Inclusion Criteria:

* Good oral hygiene with compliance to perform strict oral hygiene measures (periodontal screening index 0-1).
* Slight malposition.
* Teeth with spacing.
* Teeth with discoloration

Exclusion Criteria:

* Advanced periodontitis, gingivitis, or recession.
* Abutments with subgingival restorations or root caries.
* Parafunctional habits.
* Undergoing orthodontic treatment.
* Presence of orthodontic appliance.
* Obvious dentition malalignment.
* Mandibular prognathism.
* Maxillary retrognathism.
* Smokers.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Color stability assessment | up to 12 months
  VITA Easyshade® Advance spectrophotometer will be used to measure the shade on the CIELab system, which defines color on 3 axes: L*, lightness, ranging from 0 (black) to 100 (white); and a* and b*, chromatic characteristics ranging from red (+a*) to green (-a*) and yellow (+b*) to blue (-b*) The color will be measured 3 times, and the mean L*, a*, and b* values will be calculated and used to measure color change (delta E)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt